CLINICAL TRIAL: NCT00425347
Title: Phase I, Multi-Center, Open-Label, Dose Escalation Study of HuLuc63 (Humanized Anti-CS1 Monoclonal IgG1 Antibody) in Subjects With Advanced Multiple Myeloma
Brief Title: Phase I, Multi-Center, Open-Label, Dose Escalation Study of HuLuc63 in Subjects With Advanced Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Facet Biotech (Industry)
Responsible Party: Lisa Bell, Senior Director, Facet Biotech
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HuLuc63-1701; NCT00429741 (obsolete NCT alias)
Record Dates: First submitted 2007-01-18; First posted 2007-01-22 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma, MM, plasma cell myeloma, cancer
MeSH Terms: conditions — Multiple Myeloma; Neoplasms | interventions — elotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: HuLuc63 — Not applicable for HuLuc63.

SUMMARY:
To identify the MTD of HuLuc63 administered intravenously (IV) for 4 doses.2. To evaluate the safety of HuLuc63 IV given every other week for 4 doses.

ELIGIBILITY:
Inclusion Criteria:

Eligible subjects will be considered for inclusion in this study if they meet all of the following criteria:

* Males or females, age 18 years or older.
* Diagnosis of advanced multiple myeloma, after at least 2 prior therapies for MM.
* Measurable disease M component in serum (at least 0.5 G/dL) and/or urine (≥0.2 g excreted in a 24-hour collection sample).
* Not eligible for stem cell or bone marrow transplant or have refused stem cell or bone marrow transplant or have relapsed after autologous or allogeneic stem cell or bone marrow transplant.
* ECOG performance status 0-2 (Appendix E).
* ALT or AST ≤3 x ULN.
* Total bilirubin ≤2 x ULN (unless related to MM).
* Serum creatinine ≤2.0 mg/dL (unless related to MM, then ≤ 3.0 mg/dL).
* Must have adequate bone marrow function defined as: Absolute neutrophil count >1,000 cells/mm3; platelets ≥75,000 cells/mm3; and hemoglobin ≥8 g/dL. No platelet transfusion within 72 hours of obtaining screening platelet count.
* Serum calcium (corrected for albumin) level within normal range (treatment of hypercalcemia is allowed and subject may enroll if hypercalcemia returns to normal with treatment).
* Signed and dated informed consent.
* Use of appropriate contraception where applicable.
* Negative pregnancy test within 48 hours prior to first dose in women of childbearing potential.
* Must have 2-dimensional echocardiogram or MUGA indicating LVEF ≥ 45% within 30 days prior to first dose of study drug.
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local subject privacy regulations).

Exclusion Criteria:

Subjects will be ineligible for this study if they meet any one of the following criteria:

* Life expectancy of less than 3 months.
* Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease-free for at least 5 years.
* Plasma cell leukemia (active or prior).
* Uncontrolled medical problems such as diabetes mellitus, coronary artery disease, hypertension, unstable angina, arrhythmias, pulmonary, hepatic, and renal diseases unless renal insufficiency is felt to be secondary to multiple myeloma (serum creatinine > 2.0 mg/dL).
* Solitary bone or solitary extramedullary plasmacytoma as the only evidence of plasma cell dyscrasia.
* Corticosteroid, Velcade® or other proteosome inhibitor, thalidomide, lenalidomide (Revlimid®), or melphalan within 2 weeks of the first dose of HuLuc63; nitrogen mustard agents within 6 weeks of the first dose of HuLuc63.
* Investigational drug within 4 weeks or 5 half-lives (whichever is greater) of the first dose of HuLuc63.
* Stem cell or bone marrow transplant within 12 weeks prior to the first dose of HuLuc63.
* Biological agents including intravenous immune globulin (IVIG) and monoclonal antibodies within 4 weeks of the first dose of HuLuc63.
* Neuropathy >Grade 2 (according to the NCI CTCAE v3.0 criteria scale).
* Symptomatic orthostatic hypotension.
* Evidence of amyloidosis.
* Known active infections requiring antibiotics, antivirals, or antifungals.
* Serious psychiatric illness, active alcoholism, or drug addiction that may hinder or confuse follow-up evaluation.
* Hypersensitivity to recombinant proteins or excipients in the investigational agent.
* Any condition that in the investigator's opinion makes the subject unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-12; Primary Completion 2008-08 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Not applicable for this trial. | Not applicable for this trial.

CONTACTS AND LOCATIONS:
Overall Officials: William Bensinger, MD, Principal Investigator — Fred Hutchinson Cancer Center; Robert Dean, MD, Principal Investigator — The Cleveland Clinic; Frits van Rhee, M.D., Principal Investigator — Arkansas Cancer Research Center; Seema Singhal, M.D., Principal Investigator — Northwestern University Feinberg School of Medicine; Jeffrey A. Zonder, M.D., Principal Investigator — Wayne State University; Samer Al-Homsi, M.D., Principal Investigator — University of Massachusetts Memorial Healthcare; Nikhil Munshi, M.D., Principal Investigator — Dana-Farber Cancer Institute; Ann Mohrbacher, M.D., Principal Investigator — USC/Norris Cancer Hospital
Locations (8):
- United States (8):
  - Arkansas Cancer Research Center, Little Rock, Arkansas
  - USC/Norris Cancer Hospital, Los Angeles, California
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Healthcare- Univ. Campus, Worcester, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Cleveland Clinic, Cleveland, Ohio
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- See also: Related Info — http://www.facetbiotech.com